CLINICAL TRIAL: NCT02322229
Title: Assessment of Anatomical and Functional Outcomes in Subjects Treated With Ocriplasmin for Vitreomacular Traction/Symptomatic Vitreomacular Adhesion (VMT/sVMA)
Brief Title: Ocriplasmin for Vitreomacular Traction/Symptomatic Vitreomacular Adhesion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTA255-P001
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2017-10

CONDITIONS: Vitreomacular Traction; Vitreomacular Adhesion
Keywords: VMT; sVMA; vitrectomy; ocriplasmin
MeSH Terms: interventions — microplasmin; Plasminogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ocriplasmin (Experimental): Ocriplasmin 0.125 mg in a 0.1 mL volume administered as a single dose by intravitreal (IVT) injection
  Interventions: Drug: Ocriplasmin 0.125 mg in a 0.1 mL volume

INTERVENTIONS:
Drug: Ocriplasmin 0.125 mg in a 0.1 mL volume
  Other Names: JETREA™®

SUMMARY:
The purpose of this study is to observe the anatomical and functional outcomes of ocriplasmin (JETREA™®) over a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of VMT/sVMA, with evidence of focal VMT visible on Spectral Domain - Optical Coherence Tomography (SD-OCT).
* Read, sign, and date an Institutional Review Board/Ethics Committee-approved informed consent form.
* Willing and able to attend all study visits.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, test positive on a urine pregnancy test, intend to become pregnant during the study period, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Hypersensitivity to ocriplasmin or any of the JETREA™® excipients.
* Active or suspected intraocular or periocular infection in either eye.
* Participation in any interventional clinical trial within 30 days prior to baseline.
* Presence of epiretinal membrane (ERM) over the macula at baseline in the study eye.
* Broad VMT/VMA > 1500 microns at baseline in the study eye.
* History of vitrectomy in the study eye.
* History of laser photocoagulation to the macula in the study eye.
* Any relevant concomitant ocular condition in the study eye that, in the opinion of the Investigator, could be expected to worsen or require surgical intervention during the study period.
* Macular hole of > 400 microns diameter in the study eye.
* High myopia in the study eye.
* Pseudo-exfoliation, Marfan's syndrome, phacodonesis, or any other finding in the study eye that, in the Investigator's opinion, suggests lens/zonular instability.
* Aphakia in the study eye.
* History of retinal detachment in the study eye.
* Recent ocular surgery or ocular injection in the study eye within the past 90 days (including laser therapy).
* Proliferative diabetic retinopathy or ischemic retinopathies in the study eye.
* Retinal vein occlusions in the study eye.
* Exudative age-related macular degeneration (AMD) in the study eye.
* Vitreous hemorrhage in the study eye.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Dir of Operations, Ophthalmology, GMA, Study Director — Alcon, A Novartis Division
Locations (1):
- Contact Alcon Laboratories (Australia) for Trial Locations, New South Wales, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 sites located in Australia and 1 site located in New Zealand.
Pre-assignment Details: Of the 62 enrolled, 10 subjects were exited as screen failures prior to initiation of treatment. This reporting group includes all eligible subjects (52).
Period: Overall Study
Arm/Group | Ocriplasmin
Started | 52
Completed | 50
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who received treatment with investigational product (IP) and had at least 1 post-treatment measurement of SD-OCT (Full Analysis Set).
Groups:
- Ocriplasmin: Ocriplasmin 0.125 mg in a 0.1 mL volume administered as a single dose by IVT injection
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Non-surgical Resolution of Focal VMT/sVMA at Day 28, as Determined by Central Reading Center (CRC) Spectral Domain Optical Coherence Tomography (SD-OCT) Evaluation
Description: Vitreous separation was assessed, by SD-OCT according to CRC OCT image reading, into 1 of 12 categories, where the targeted status of VMA resolution was 7=Vitreous attached only at optic nerve (ON) or at ON and elsewhere, but not attached in macular, 9=Vitreous visible with complete separation and no attachment, and 10=No visible vitreous separation, which needed to be reached without prior vitrectomy. The assessment of resolution of VMT/sVMA was based upon the anatomical resolution of VMA only, i.e. no resolution of the related symptoms was considered. One eye (study eye) contributed to the analysis.
Time Frame: Day 28
Population: Full Analysis Set. Missing data imputed using the last observation carried forward (LOCF) method. Subjects who had vitrectomy after VMA resolution are considered as 'no VMA resolution' after timepoint of vitrectomy.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 52
percentage of subjects | 26.9

2. Secondary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) at Distance at Days 7, 28, 90, and 180
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) testing. BCVA was determined as follows: if tested at 4 meters, BCVA=the number of letters read correctly at 4 meters+30; if tested at 1 meter, BCVA=the number of letters read correctly at 1 meter, with 83-84 representing normal vision. BCVA change was defined as a change in letters read from the baseline assessment. A positive change value indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 7, Day 28, Day 90, Day 180
Population: Full Analysis Set. Missing data imputed using the LOCF method. BCVA values after a vitrectomy are imputed with the last non-missing value prior to the vitrectomy.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 52
letters
  Baseline (BL) | 70.6 (10.62)
  Change from BL at Day 7 | -1.8 (7.09)
  Change from BL at Day 28 | 1.0 (7.67)
  Change from BL at Day 90 | 2.1 (8.07)
  Change from BL at Day 180 | 3.3 (9.16)

3. Secondary Outcome: Percentage of Subjects With Closure of Macular Hole (MH), at Days 7, 28, 90, and 180 (if Present at Baseline)
Description: The closure of macular hole (a full thickness defect of the retinal tissue involving the anatomical fovea) is defined as a flattened and reattached hole rim along the whole circumference of macular hole. Closure was determined by SD-OCT evaluation and the percentage of subjects tabulated. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 28, Day 90, Day 180
Population: This analysis population includes all subjects in Full Analysis Set with MH at baseline (n=4). Subjects who had vitrectomy after MH closure are considered as 'no MH closure' after the timepoint of vitrectomy.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 4
percentage of subjects
  Day 7 | 25.0
  Day 28 | 50.0
  Day 90 | 50.0
  Day 180 | 50.0

4. Secondary Outcome: Percentage of Subjects With Non-surgical Resolution of VMT/sVMA at Days 7, 90, and 180
Description: As described in Primary Outcome Measure
Time Frame: Baseline (Day 0), Day 7, Day 90, Day 180
Population: Full Analysis Set. Missing data imputed for Days 90 and 180 using the LOCF method. Subjects who had vitrectomy are considered as 'no VMA resolution' after the timepoint of vitrectomy.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 52
percentage of subjects
  Day 7 | 19.2
  Day 90 | 38.5
  Day 180 | 40.4

5. Secondary Outcome: Percentage of Subjects Experiencing Pars Plana Vitrectomy (PPV) at Day 180
Description: Pars plana vitrectomy (the surgical removal of vitreous gel from the eye) was captured in Concomitant Ocular Procedures. One eye (study eye) contributed to the analysis.
Time Frame: Day 180
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 52
percentage of subjects | 7.7

6. Secondary Outcome: Change From Baseline in Central Foveal Thickness at Days 28 and 180
Description: Central foveal thickness (CFT) was determined by subtracting the measurements in subretinal fluid (SRF) and retinal pigment epithelium (RPE) elevation and/or subretinal hyper-reflective material (SHRM) from the value in total retinal measurement. The change was defined as a change from baseline values of CFT. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 28, Day 180
Population: Missing data is imputed using the LOCF method. CFT values after a vitrectomy are imputed with the last non-missing value prior to the vitrectomy.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 52
Microns
  Baseline (BL) | 302.3 (161.23)
  Change from BL at Day 28 | -35.5 (95.53)
  Change from BL at Day 180 | -17.6 (143.63)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 7 months). AEs are reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment (ie, initiation of treatment with test article) regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- Jetrea: Subjects exposed to Ocriplasmin 0.125 mg in a 0.1 mL volume administered as a single dose by IVT injection
Arm/Group | Pretreatment | Jetrea
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/62 | 5/52
Other Adverse Events (participants affected / at risk) | 1/62 | 41/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=62) | Jetrea (N=52)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Macular hole (Eye disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=62) | Jetrea (N=52)
Eye pain (Eye disorders) | 0 | 4
Lacrimation increased (Eye disorders) | 0 | 3
Metamorphopsia (Eye disorders) | 0 | 8
Photopsia (Eye disorders) | 0 | 27
Vision blurred (Eye disorders) | 0 | 12
Visual acuity reduced (Eye disorders) | 0 | 11
Visual impairment (Eye disorders) | 0 | 9
Vitreous floaters (Eye disorders) | 1 | 6
Influenza (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.